CLINICAL TRIAL: NCT00820664
Title: A Randomized Clinical Trial to Evaluate the Effects of Estrogen on Uterine Endometrium in Healthy Postmenopausal Women
Brief Title: A Clinical Study to Evaluate the Effects of Estrogen in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-122; 2009_505
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Results first posted 2010-05-07 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Postmenopausal Symptoms
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 17β-estradiol 2.0 milligrams (Active Comparator): Estrace 2.0 mg tablet
  Interventions: Drug: Comparator: Estrace 2 mg
- 17β-estradiol 0.5 milligrams (Active Comparator): Estrace 0.5 mg tablet
  Interventions: Drug: Comparator: Estrace 0.5 mg
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: Estrace 0.5 mg — 0.5 mg tablet taken once daily for 28 days
  Other Names: Estrace
  Arms: 17β-estradiol 0.5 milligrams
Drug: Comparator: Estrace 2 mg — 2 mg tablets taken once daily for 28 days.
  Other Names: Estrace
  Arms: 17β-estradiol 2.0 milligrams
Drug: Comparator: Placebo — Placebo 0 mg capsule taken once daily for 28 days
  Arms: 3

SUMMARY:
The purpose of this study is to examine the effect of two different dose levels of estrogen or placebo in healthy postmenopausal women by measuring the changes in hormone levels and examining the changes in the uterine lining (endometrium).

ELIGIBILITY:
Inclusion Criteria:

* Patient is a healthy postmenopausal woman less than or equal to 65 years of age with onset of menopause less than or equal to 10 years prior to prestudy visit 1
* Patient has a uterus and no history of uterine bleeding in the past 3 months
* Patient has not had a previous endometrial biopsy within the last 4 weeks
* Patient has had a normal mammogram within the last 11 months
* Patient has had a normal pap-smear within the past 3 years prior to screening
* Patient has had a normal transvaginal ultrasound of the endometrium
* Patient is willing to avoid strenuous physical activity such as strenuous or unaccustomed weight lifting, running, bicycling, etc for the duration of the study
* Patient agrees to not consume grapefruit products beginning approximately 2 weeks prior to the first dose of study drug and throughout the study
* Patient agrees to limit daily consumption of alcohol. During the study, daily alcohol consumption should not be more than 2 glasses
* Patient agrees to limit daily consumption of caffeine. During the study, daily caffeine consumption should not exceed 3 cups of coffee
* Patient is a non-smoker

Exclusion Criteria:

* Patient is mentally or legally incapacitated
* Patient has a history of any first degree relatives with breast or endometrial cancer
* Patient has a history of multiple and/or severe allergies to prescription or non-prescription drugs or food
* Patient has used any type of estrogen or progesterone preparation unless followed by appropriate wash-out periods
* Patient has had surgery, donated approximately 500 mL of blood or has participated in another investigational study within the last 4 weeks
* Patient has a history of deep vein thromboses, coronary artery disease, heart attack or stroke
* Patient is a current user of illegal drugs
* Patient has a history of hypersensitivity to estrogen products
* Patient is unable to refrain from using anti-coagulants

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited through advertisement and review of patient databases at Comprehensive Phase I, USA, between December 2008 and April 2009.
Pre-assignment Details: Major entry criteria - healthy postmenopausal women within 10 years of attaining menopause as determined by follicle-stimulating hormone (FSH) and estradiol levels within range of postmenopause, and other criteria. Normal transvaginal ultrasound at screening with endometrial thickening at < 5.0 mm.
Period: Overall Study
Arm/Group | 17β-estradiol 2.0 Milligrams | 17β-estradiol 0.5 Milligrams | Placebo
Started | 9 | 11 | 9
Completed | 9 | 11 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 17β-estradiol 2.0 Milligrams | 17β-estradiol 0.5 Milligrams | Placebo | Total
Number analyzed (Participants) | 9 | 11 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.11 (3.76) | 53.91 (5.65) | 55.33 (3.04) | 54.41 (4.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 9 | 29
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 1 | 0 | 0 | 1
  White | 8 | 11 | 9 | 28
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.87 (3.95) | 28.69 (2.74) | 27.43 (1.98) | 28.05 (2.92)

OUTCOME MEASURES:

1. Primary Outcome: Immunohistochemistry (IHC) Proliferative Effects Measurement
Description: Ratio of the total number of positively stained cell nuclei to the total number of cell nuclei. Proliferating endometrial cells express the Ki-67 antigen. The ratio was converted to a percent proliferating cells by taking the number of Ki-67 positive stained nuclei in a given field and dividing by the total number of nuclei in that field and multiplying by 100. At least 5 high power fields were scored in this manner and an aggregate percent Ki-67 positive cells was reported. Square root transformation was taken to make it approximately normally distributed for an ANOVA model to apply.
Time Frame: 4 weeks
Population: Though 29 subjects were enrolled, only 20 subjects had biopsy samples that were deemed adequate for Ki-67 immunohistochemical analysis at Week 4.
Measure: Least Squares Mean (95% Confidence Interval); unit: Square root of % positive stained cells
Arm/Group | 17β-estradiol 2.0 Milligrams | 17β-estradiol 0.5 Milligrams | Placebo
Number analyzed (Participants) | 6 | 8 | 6
Square root of % positive stained cells | 0.73 [0.61 to 0.86] | 0.43 [0.32 to 0.54] | 0.25 [0.12 to 0.37]
Statistical Analysis 1: Comparison: 17β-estradiol 2.0 Milligrams vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — 1-sided, alpha=0.05; A one-way ANOVA model with term treatment was fit to the square root transformed response; Least Squares Mean = 0.49, 95% CI [0.31 to 1.00]
Statistical Analysis 2: Comparison: 17β-estradiol 0.5 Milligrams vs Placebo; Test type: Superiority or Other; p = 0.032, ANOVA — 1-sided, alpha=0.05; A one-way ANOVA model with term treatment was fit to the square root transformed response; Least Squares Mean = 0.19, 95% CI [0.02 to 1.00]

2. Secondary Outcome: Mean Gene Expression Intensity After 4 Weeks of Either 0.5 or 2 mg Estrace Compared to Placebo.
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Reported AE data were collected during the period of the study from date of informed consent to the 14 day follow up period following completion of treatment.
Description: Clinical staff telephoned subjects daily during the study, in between clinic visits and asked the subjects if they had experienced any adverse experiences.
Arm/Group | 17β-estradiol 2.0 Milligrams | 17β-estradiol 0.5 Milligrams | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 7/9 | 6/11 | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 17β-estradiol 2.0 Milligrams (N=9) | 17β-estradiol 0.5 Milligrams (N=11) | Placebo (N=9)
Vision Blurred (Eye disorders) | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1 | 0
Feeling Cold (General disorders) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1
Headache (Nervous system disorders) | 2 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 4 | 1 | 0
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The registered secondary outcome: "Mean gene expression intensity after 4 weeks of either 0.5 or 2 mg Estrace compared to placebo" results are not available because of inadequate quantity and quality of tissue samples that were obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.